CLINICAL TRIAL: NCT03936959
Title: A Phase 1 Study of LY3434172, a Bispecific Antibody Monotherapy in Advanced Solid Tumors
Brief Title: A Study of LY3434172, a PD-1 and PD-L1 Bispecific Antibody, in Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study did not achieve its primary objective due to early termination of the study
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17101; J1E-MC-JZEA (Other: Eli Lilly and Company); 2018-003871-37 (EudraCT Number)
Record Dates: First submitted 2019-04-26; First posted 2019-05-03 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Advanced Cancer
Keywords: PD-1; PD-L1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 3 Milligram (mg) - 10 mg LY3434172 (Experimental): 3 mg LY3434172 administered intravenously (IV) on Day 1 Cycle 1 of 28-day cycle. 10 mg LY3434172 administered IV on Day 15 Cycle 1 of 28-day cycle.
  Participants continued to receive study treatment until they met a criterion for discontinuation.
  Interventions: Drug: LY3434172
- 30 mg LY3434172 (Experimental): 30 mg LY3434172 administered IV on Day 1 and Day 15 of 28-day cycle. Participants continued to receive study treatment until they met a criterion for discontinuation.
  Interventions: Drug: LY3434172
- 100 mg LY3434172 (Experimental): 100 mg LY3434172 administered IV on Day 1 and Day 15 of 28-day cycle. Participants continued to receive study treatment until they met a criterion for discontinuation.
  Interventions: Drug: LY3434172

INTERVENTIONS:
Drug: LY3434172 — Administered IV

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of the study drug LY3434172, a PD-1/PD-L1 bispecific antibody, in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Must have histological or cytological evidence of a diagnosis of cancer that is not amenable/resistant to approved standard-of-care therapy for the following solid tumors: Melanoma, non-small cell lung cancer (NSCLC), squamous cell carcinoma of the head and neck (SCCHN), urothelial cancer, gastric cancer, colorectal cancer, biliary tract cancer, anal cancer, nasopharyngeal cancer, esophageal cancer, SCLC, ovarian cancer, mesothelioma, pan-tumor MSIhi solid tumors, hepatocellular carcinoma, merkel cell cancer, cutaneous squamous cell carcinoma, endometrial cancer, breast cancer, cervical cancer, thyroid cancer, salivary cancer, and prostate cancer who have received at least one line of standard systemic therapy for their respective tumor type in the metastatic setting with progressive locally advanced or metastatic disease. Prior anti-programmed death 1 (PD-1) and anti-programmed death ligand 1 (PD-L1) allowed if they received another therapy immediately prior to this study or there has been a lapse of approximately ≥90 days from prior therapy.
* Must be willing to undergo pretreatment and on-treatment core needle or excisional tumor biopsies.
* Have at least one measurable lesion assessable as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Have adequate organ function.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have an estimated life expectancy of 12 weeks, in the judgment of the investigator.

Exclusion Criteria:

* Have symptomatic central nervous system (CNS) malignancy or metastasis not requiring concurrent treatment, including but not limited to surgery, radiation, corticosteroids and/or anticonvulsants to treat CNS metastases, and their disease is asymptomatic and radiographically stable for at least 30 days.
* Have moderate or severe cardiovascular disease.
* Have active or suspected autoimmune disease (eg. autoimmune vasculitis, autoimmune myocarditis, among others).
* Have serious concomitant systemic disorder that would compromise the participant's ability to adhere to the protocol, including known infection with human immunodeficiency virus (HIV) unless they are well controlled on highly active antiretroviral therapy (HAART) therapy with no evidence of acquired immune deficiency syndrome (AIDS)-defining opportunistic infections within the last 2 years, and CD4 T-cells count > 350 cells/µl , active hepatitis B virus (HBV), active hepatitis C virus (HCV), active autoimmune disorders, or prior documented severe autoimmune or inflammatory disorders requiring immunosuppressive treatment.

  * Use of escalating or chronic supraphysiologic doses of corticosteroids or immunosuppressive agents (such as, exceeding 10 milligrams/day of prednisone or equivalent). Use of topical, ophthalmic, inhaled, and intranasal corticosteroids permitted.
* Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection, Crohn's disease, ulcerative colitis, or chronic diarrhea.
* Evidence of interstitial lung disease or noninfectious pneumonitis (active or treated by corticosteroid therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- St Vincent's Hospital, Sydney, New South Wales, Australia
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Institut Claudius Regaud - IUCT Oncopole, Toulouse, France
- Asan Medical Center, Songpa-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3434172, a PD-1 and PD-L1 Bispecific Antibody, in Advanced Cancer — https://trials.lillytrialguide.com/en-US/trial/1aYuXmPG4pbGQPqjXu8y8C

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers are defined as participants who were observed for both primary and secondary outcomes.
Period: Overall Study
Arm/Group | 3 Milligram (mg) - 10 mg LY3434172 | 30 mg LY3434172 | 100 mg LY3434172
Started | 3 | 4 | 3
Received at Least One Dose of Study Drug | 3 | 4 | 3
Completed | 3 | 4 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received any quantity of LY3434172, regardless of their eligibility for the study.
Groups:
- 3 mg - 10 mg LY3434172: 3 mg LY3434172 administered IV on Day 1 Cycle 1 of 28-day cycle. 10 mg LY3434172 administered IV on Day 15 Cycle 1 of 28-day cycle. Participants continued to receive study treatment until they met a criterion for discontinuation.
- Total: Total of all reporting groups
Arm/Group | 3 mg - 10 mg LY3434172 | 30 mg LY3434172 | 100 mg LY3434172 | Total
Number analyzed (Participants) | 3 | 4 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 1 | 5
  >=65 years | 2 | 1 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 6
  Male | 1 | 1 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 2 | 3 | 1 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 0 | 0 | 1 | 1
  Belgium | 1 | 1 | 1 | 3
  United States | 2 | 3 | 0 | 5
  Australia | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT is defined as adverse event/s of grade 3 or higher that occurs during the DLT observation period, which is Cycle 1 of each dose escalation cohort, and is clinically significant and definitely, probably, or possibly related to LY3434172, in the opinion of the investigator.
Time Frame: Baseline through Cycle 1 (Up to 42 Day Cycle)
Population: All participants who received any quantity of LY3434172, regardless of their eligibility for the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg - 10 mg LY3434172 | 30 mg LY3434172 | 100 mg LY3434172
Number analyzed (Participants) | 3 | 4 | 3
Participants | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of LY3434172
Description: PK: Cmin of LY3434172
Time Frame: PK: Cycle 1 Day 1 (C1D1): Predose; 1 hour(h); 3 h; 24 h; 72 h; 168 h post-infusion; Cycle 1 Day 15 (C1D15): Predose; 1 h; 3 h; 24 h; 72 h; 168 h post-infusion
Population: All participants who received at least one dose of LY3434172 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- 3 mg - 10 mg LY3434172: 3 mg LY3434172 administered intravenously (IV) on Day 1 Cycle 1 of 28-day cycle. 10 mg LY3434172 administered IV on Day 15 Cycle 1 of 28-day cycle. Participants continued to receive study treatment until they met a criterion for discontinuation.
Arm/Group | 3 mg - 10 mg LY3434172 | 30 mg LY3434172 | 100 mg LY3434172
Number analyzed (Participants) | 3 | 4 | 3
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | NA (NA) — Cmin non calculable, value is less than lower limit of quantification (<LLOQ). | 775 (107) | 4150 (254)
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 3 | 3
  Cycle 1 Day 15 | NA (NA) — Cmin non calculable, value is <LLOQ. | 1017 (63) | 5600 (85)

3. Secondary Outcome: PK: Maximum Concentration (Cmax) of LY3434172
Description: PK: Cmax of LY3434172
Time Frame: PK: Cycle 1 Day 1 (C1D1): Predose; 1 hour(h); 3 h; 24 h; 72 h; 168 h post-infusion; C1D15: Predose; 1 h; 3 h; 24 h; 72 h; 168 h post-infusion
Population: All participants who received at least one dose of LY3434172 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 3 mg - 10 mg LY3434172 | 30 mg LY3434172 | 100 mg LY3434172
Number analyzed (Participants) | 3 | 4 | 3
ng/mL
  Cycle 1 Day 1 | 734 (19.1) | 8250 (17.7) | 22700 (60.8)
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 4 | 3
  Cycle 1 Day 15 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation (CV) non calculable, individual PK parameters reported: 834 ng/mL; 2280 ng/mL | 18600 (52.9) | 43000 (58.5)

4. Secondary Outcome: PK: Area Under the Curve From Zero to Time to Last Measurable Concentration (AUC0-tlast) of LY3434172
Description: PK: AUC 0-tlast of LY3434172
Time Frame: as for outcome 3
Population: All participants who received at least one dose of LY3434172 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | 3 mg - 10 mg LY3434172 | 30 mg LY3434172 | 100 mg LY3434172
Number analyzed (Participants) | 3 | 4 | 3
hour*nanogram per milliliter (hr*ng/mL)
  C1D1 | 7280 (51.0) | 584000 (31.5) | 1900000 (121)
  C1D15: number analyzed (Participants) | 2 | 3 | 3
  C1D15 | NA (NA) — Geometric Mean and CV non calculable, individual PK parameters reported: 9770 hr*ng/mL; 29600 hr*ng/mL. | 559000 (239) | 3010000 (19.9)

5. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With a Complete Response (CR) or Partial Response (PR)
Description: ORR: Percentage of participants who have received any amount of study drug, have at least one postbaseline tumor image, and achieved a best overall response (BOR) of confirmed Complete Response (CR) is defined a disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). Partial Response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline through Measured Progressive Disease (Up to 8.4 Months)
Population: All participants who received any quantity of LY3434172, regardless of their eligibility for the study.
Measure: Number; unit: Percentage of participants
Arm/Group | 3 mg - 10 mg LY3434172 | 30 mg LY3434172 | 100 mg LY3434172
Number analyzed (Participants) | 3 | 4 | 3
Percentage of participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 33.3

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined only for responders (participants with a confirmed CR or PR). It is measured from the date of first evidence of a confirmed CR or PR to the date of the first observed radiographically documented progressive disease (PD), or the date of death due to any cause, whichever is earlier. If a responder is not known to have died or have objective progression as of the data inclusion cutoff date, DoR will be censored at the date of the last complete objective progression-free disease assessment.
Time Frame: Date of CR or PR to Date of Objective Progression or Death Due to Any Cause (Up to 8.4 Months)
Population: All participants who received any quantity of LY3434172, regardless of their eligibility for the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 3 mg - 10 mg LY3434172 | 30 mg LY3434172 | 100 mg LY3434172
Number analyzed (Participants) | 0 | 0 | 1
Months |  |  | NA [NA to NA] — Median and 95% Confidence interval could not be calculated as there was only one participant. Individual value reported: 1.9 months, (57 days). DoR censored at the last available scan prior to data cut-off.

7. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the time from the date of first study treatment until the first evidence of confirmed CR or PR.
Time Frame: Baseline to Date of CR or PR (Up to 8.4 Months)
Population: All participants who received any quantity of LY3434172, regardless of their eligibility for the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 3 mg - 10 mg LY3434172 | 30 mg LY3434172 | 100 mg LY3434172
Number analyzed (Participants) | 0 | 0 | 1
Months |  |  | NA [NA to NA] — Median and 95% Confidence interval could not be calculated as there was only one participant. Individual value reported: 1.7 months (52 days).

8. Secondary Outcome: Disease Control Rate (DCR): Percentage of Participants Who Exhibit Stable Disease (SD), CR or PR
Description: Disease control rate is defined as the number of participants with SD, confirmed PR, or confirmed CR (CR+PR+SD) divided by the number of enrolled participants who have received any quantity of study treatment.
Time Frame: Baseline through Measured Progressive Disease (Up to 8.4 Months)
Population: All participants who received any quantity of LY3434172, regardless of their eligibility for the study.
Measure: Number; unit: percentage of participants
Arm/Group | 3 mg - 10 mg LY3434172 | 30 mg LY3434172 | 100 mg LY3434172
Number analyzed (Participants) | 3 | 4 | 3
percentage of participants | 66.7 | 25.0 | 66.7

ADVERSE EVENTS:
Time Frame: Baseline Up to 16.7 Months
Description: All participants who received any quantity of LY3434172, regardless of their eligibility for the study.
Groups:
- 3 mg -10 mg LY3434172: 3 mg LY3434172 administered IV on Day 1 Cycle 1 of 28-day cycle. 10 mg LY3434172 administered IV on Day 15 Cycle 1 of 28-day cycle. Participants continued to receive study treatment until they met a criterion for discontinuation.
Arm/Group | 3 mg -10 mg LY3434172 | 30 mg LY3434172 | 100 mg LY3434172
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/4 | 2/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg -10 mg LY3434172 (N=3) | 30 mg LY3434172 (N=4) | 100 mg LY3434172 (N=3)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg -10 mg LY3434172 (N=3) | 30 mg LY3434172 (N=4) | 100 mg LY3434172 (N=3)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (7) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (5) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 2 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated by sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT03936959/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT03936959/SAP_001.pdf